CLINICAL TRIAL: NCT03852719
Title: A Multicenter, Open-label, Randomized Phase 3 Clinical Study to Assess Efficacy and Safety of Bulevirtide in Patients With Chronic Hepatitis Delta
Brief Title: Study to Assess Efficacy and Safety of Bulevirtide in Participants With Chronic Hepatitis Delta (CHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MYR301; 2019-001213-17 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-02-25 (Actual); Results first posted 2022-10-28 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Chronic Hepatitis Delta
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — bulevirtide; myrcludex-B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Delayed Treatment/Bulevirtide 10 mg/day (Experimental): After an observational period of 48 weeks, participants will receive treatment with bulevirtide 10 mg/day subcutaneously (SC) for 96 weeks and will be followed for up to 96 weeks (Up to Week 240).
  Interventions: Drug: Bulevirtide
- Bulevirtide 2 mg/day (Experimental): Participants will receive bulevirtide 2 mg/day SC for 144 weeks and will be followed for up to 96 weeks (Up to Week 240).
  Interventions: Drug: Bulevirtide
- Bulevirtide 10 mg/day (Experimental): Participants will receive bulevirtide 10 mg/day SC for 144 weeks and will be followed for up to 96 weeks (Up to Week 240).
  Interventions: Drug: Bulevirtide

INTERVENTIONS:
Drug: Bulevirtide — Administered via SC injections
  Other Names: Myrcludex B; Hepcludex®

SUMMARY:
The primary objective of this study is to evaluate the efficacy of bulevirtide administered subcutaneously (SC) for 48 weeks at a dose of 2 mg or 10 mg once daily for treatment of chronic hepatitis delta (CHD) in comparison to delayed treatment.

The main goal of this study is to determine the effectiveness of bulevirtide in participants randomized to bulevirtide 2 mg or 10 mg once daily SC as compared to participants randomized to delayed treatment for 48 weeks. Treatment will continue through Week 144 (participants randomized to delayed treatment will change to bulevirtide 10 mg once daily SC after Week 48 through Week 144). All participants will be followed off-treatment for an additional 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Positive serum anti-hepatitis delta virus (HDV) antibody results or polymerase chain reaction (PCR) results for serum/ plasma HDV ribonucleic acid (RNA) for at least 6 months before screening.
3. Positive PCR results for serum/plasma HDV RNA at screening.
4. Alanine transaminase level > 1 x upper limit of normal (ULN), but less than 10 x ULN.
5. Serum albumin > 28 g/L.
6. Negative urine pregnancy test for females of childbearing potential.
7. Inclusion criteria for females:

   * Postmenopausal for at least 2 years, or
   * Surgically sterile (total hysterectomy or bilateral oophorectomy, bilateral tubal ligation, staples, or another type of sterilization), or
   * Abstinence from heterosexual intercourse throughout the study, or
   * Willingness to use highly effective contraception (double barrier method or barrier contraception in combination with hormonal or intrauterine contraceptive) throughout the study and for 3 months after the last dose of the study medication for individuals discontinued during the treatment period.
8. Individuals must agree to use a highly effective contraception (double barrier method or barrier contraception in combination with hormonal or intrauterine contraceptive used by female partners) and not to donate sperm throughout the study and for 3 months after the last dose of the study medication for individuals discontinued during the treatment period.

Exclusion Criteria:

1. Child-Pugh hepatic insufficiency score over 7 points. Uncomplicated oesophageal varices allowed; Individuals with current bleeding or ligation, or history of bleeding or ligation within the last 2 years are excluded.
2. Hepatitis C virus (HCV) or uncontrolled human immunodeficiency virus (HIV) coinfection. Individuals with HCV antibodies can be enrolled, if screening HCV RNA test is negative. Individuals with HIV infection can be enrolled if cluster of differentiation (CD4+) cell counts are >500/mL and HIV RNA is below limit of detection for at least 12 months.
3. Creatinine clearance < 60 mL/min as estimated using Cockcroft-Gault formula.
4. Total bilirubin ≥ 34.2 µmol/L. (Individuals with higher total bilirubin values may be included after the consultation with the Study Medical Monitor, if such elevation can be clearly attributed to Gilbert's syndrome associated with low-grade hyperbilirubinemia.)
5. Evidence of an active or suspected malignancy or a history of malignancy, or an untreated pre-malignancy disorder within the last 5 years (with the exception of successfully treated carcinoma of the cervix in situ and successfully treated basal cell carcinoma and squamous cell carcinoma not less than 1 year prior to screening [and no more than 3 excised skin cancer within the last 5 years prior to screening]) or history of hepatic carcinoma.
6. Systemic connective tissue disorders.
7. New York Heart Association (NYHA) class III-IV congestive heart failure.
8. Individuals with uncontrolled arterial hypertension: systolic blood pressure > 150 mm Hg and/ or diastolic blood pressure > 100 mm Hg at Screening.
9. Previous or unstable concurrent diseases or conditions that prevent individual's enrolment into the study.
10. Individuals with mental disorders or social circumstances that preclude them from following protocol requirements.
11. Current or previous (within last 2 years) decompensated liver disease, including coagulopathy, hepatic encephalopathy and esophageal varices hemorrhage.
12. One or more additional known primary or secondary causes of liver disease, other than hepatitis B (e.g., alcoholism, autoimmune hepatitis, malignancy with hepatic involvement, hemochromatosis, alpha-1 antitrypsin deficiency, Wilson's Disease, other congenital or metabolic conditions affecting the liver, congestive heart failure or other severe cardiopulmonary disease, etc.). Gilbert's syndrome, a benign disorder associated with low-grade hyperbilirubinemia, will not exclude individuals from participation in this trial. Autoimmune hepatitis stigmata attributed to HDV infection in the opinion of the investigator are allowed.
13. White blood cells (WBC) count < 3000 cells/mm^3 (<1500 if African individuals).
14. Neutrophil count < 1500 cells/mm^3 (<1000 if African individuals).
15. Platelet count < 60,000 cells/mm^3.
16. Use of prohibited psychotropic agents at Screening.
17. Use of interferons within 6 months before Screening.
18. History of solid organ transplantation.
19. Current alcohol abuse or alcohol abuse within 6 months prior to enrolment in this study; past or current drug addict.
20. History of disease requiring regular use of systemic glucocorticosteroids (inhalative glucocorticosteroids are allowed) or other immunosuppressants.
21. Pregnant or breast-feeding females.
22. Participation in another clinical study with investigational drugs within 30 days prior to randomization.
23. Receipt of bulevirtide previously, e.g. in clinical trials.
24. Inability to follow protocol requirements and undergo all protocol procedures. NOTE: Individuals with medical contraindication for liver biopsy are allowed to participate in this study. Such individuals will exempt from liver biopsy requirements in this study.

Individuals receiving prohibited treatment at Screening cannot be included into the study unless this treatment is withdrawn prior to randomization.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2024-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Medical Monitor, Study Chair — Gilead Sciences
Locations (19):
- United States (2):
  - New York University School of Medicine, an administrative unit of New York University, an education corporation, New York, New York
  - Cornell University Well Madical College, New York, New York
- Germany (5):
  - Universitätsklinikum Essen (AoR), Klinik für Gastroenterologie und Hepatologie, Essen
  - Universitätsklinikum Frankfurt Medizinische Klinik 1, Frankfurt am Main
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie und Endokrinologie, Hanover
  - Heidelberg University Hospital, Departament of Gastroenterology, Infectious Diseases, Intoxication, Heidelberg
- Italy (3):
  - Division of Gastroenterology and Hepatology, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Università di Modena e Reggio Emilia- Ospedale Civile S., Modena
  - U.O. Epatologia - Azienda Ospedaliero Universitaria Pisana, Pisa
- Russia (8):
  - State Budgetary Educational Institution of Higher Professional Education "South Ural State Medical University" of the Ministry of Healthcare of the Russian Federation, Chelyabinsk
  - Specialized clinical Infectious diseases Hospital, Krasnodar
  - Federal Budget Institution of Science "Central Research Institute of Epidemiology" of The Federal Service on Customers' Rights Protection and Human Well-being Surveillance, Moscow
  - Federal State Budgetary Institution National Research Medical Center for Phthisiopulmonology and Infectious Diseases of the Ministry of Health of the Russian Federation, Moscow
  - LLC"Clinic of Modern Medicine", Moscow
  - Moscow Regional Scientific and Research Clinical Institute, Moscow
  - LLC Medical Company "Hepatolog", Samara
  - Stavropol Regional Hospital, Stavropol
- Karolinska University Hospital Huddinge, Dept of Infectious Diseases, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wedemeyer H, Aleman S, Andreone P, Blank A, Brunetto M, Bogomolov P, et al. Bulevirtide Monotherapy at Low and High Doses in Patients With Chronic Hepatitis Delta: 24 Weeks Interim Data of the Phase 3 MYR301 Study [Poster 2730]. European Association for the Study of the Liver (EASL): The Digital International Liver Congress; 2021 23-26 June.
- [Background] Wedemeyer H, Aleman S, Brunetto M, Blank A, Andreone P, Bogomolov P, et al. Efficacy and Safety of Bulevirtide Monotherapy Given at 2 mg or 10 mg Dose Level Once Daily for Treatment of Chronic Hepatitis Delta: Week 48 Primary Endpoint Results From a Phase 3 Randomized, Multicenter, Parallel Design Study [Oral Presentation 509]. EASL The International Liver Congress; 2022 22-26 June; London, UK.
- [Background] Lampertico P, Roulot D, Wedemeyer H. Bulevirtide with or without pegIFNalpha for patients with compensated chronic hepatitis delta: From clinical trials to real-world studies. J Hepatol. 2022 Nov;77(5):1422-1430. doi: 10.1016/j.jhep.2022.06.010. Epub 2022 Jun 22. PMID 35752223
- [Background] Wedemeyer H, Aleman S, Brunetto M, Blank A, Andreone P, Bogomolov P, et al. Efficacy and Safety at 96 weeks of Bulevirtide 2 mg or 10 mg Monotherapy for Chronic Hepatitis D: Results From an Interim Analysis of a Phase 3 Randomized Study. [Oral Presentation OS-068]. EASL The International Liver Congress; 2023 21-24 June; Vienna, AUS.
- [Background] Wedemeyer H, Aleman S, Brunetto MR, Blank A, Andreone P, Bogomolov P, Chulanov V, Mamonova N, Geyvandova N, Morozov V, Sagalova O, Stepanova T, Berger A, Manuilov D, Suri V, An Q, Da B, Flaherty J, Osinusi A, Liu Y, Merle U, Schulze Zur Wiesch J, Zeuzem S, Ciesek S, Cornberg M, Lampertico P; MYR 301 Study Group. A Phase 3, Randomized Trial of Bulevirtide in Chronic Hepatitis D. N Engl J Med. 2023 Jul 6;389(1):22-32. doi: 10.1056/NEJMoa2213429. Epub 2023 Jun 22. PMID 37345876
- [Background] Wedemeyer H, Aleman S, Brunetto M, Blank A, Andreone P, Bogomolov P, Chulanov V, Mamonova N, Geyvandova N, Morozov V, Sagalova O, Stepanova T, Berger A, Ciesek S, Manuilov D, Mercier RC, Da BL, Chee GM, Li M, Flaherty JF, Lau AH, Osinusi A, Schulze Zur Wiesch J, Cornberg M, Zeuzem S, Lampertico P. Bulevirtide monotherapy in patients with chronic HDV: Efficacy and safety results through week 96 from a phase III randomized trial. J Hepatol. 2024 Oct;81(4):621-629. doi: 10.1016/j.jhep.2024.05.001. Epub 2024 May 9. PMID 38734383
- [Background] Aleman S, Brunetto M, Blank A et al. Efficacy and Safety of Bulevirtide Monotherapy for Chronic Hepatitis Delta: Posttreatment Results Through 48 Weeks After the End of Treatment From an Interim Analysis of a Randomized Phase 3 Study, MYR301; The Liver Meeting, American Association for the Study of Liver Diseases; 2024 15-19 November; San Diego, USA.
- [Background] Wedemeyer H, Aleman S, Blank A et al. Final results of MYR301: A Randomised Phase 3 Study Evaluating the Efficacy and Safety of up to 144 Weeks of Bulevirtide Monotherapy For Chronic Hepatitis Delta and 96 Weeks of Posttreatment Follow-up. EASL The International Liver Congress; 2025 7-10 May, Amsterdam, Netherlands.
- [Derived] Wong RJ, Gish RG, Jacobson IM, Lim JK, Rock M, Kinyik-Merena C, Ma H, Smith N, Kim C. Impact of Double Reflex Testing and Linkage to Treatment on Clinical Outcomes of Chronic Hepatitis Delta Virus Infection in the United States. J Viral Hepat. 2026 Jan;33(1):e70119. doi: 10.1111/jvh.70119. PMID 41405233
- [Derived] Asselah T, Lampertico P, Aleman S, Bourliere M, Streinu-Cercel A, Bogomolov P, Morozov V, Stepanova T, Lazar S, Manuilov D, Mercier RC, Tseng S, Ye L, Flaherty JF, Osinusi A, Da BL, Chee GM, Lau AH, Brunetto MR, Wedemeyer H. Bulevirtide Monotherapy Is Safe and Well Tolerated in Chronic Hepatitis Delta: An Integrated Safety Analysis of Bulevirtide Clinical Trials at Week 48. Liver Int. 2025 Apr;45(4):e16174. doi: 10.1111/liv.16174. Epub 2024 Dec 8. PMID 39648559
- [Derived] Buti M, Wedemeyer H, Aleman S, Chulanov V, Morozov V, Sagalova O, Stepanova T, Gish RG, Lloyd A, Kaushik AM, Suri V, Manuilov D, Osinusi AO, Flaherty JF, Lampertico P. Patient-reported outcomes in chronic hepatitis delta: An exploratory analysis of the phase III MYR301 trial of bulevirtide. J Hepatol. 2025 Jan;82(1):28-36. doi: 10.1016/j.jhep.2024.06.031. Epub 2024 Jul 14. PMID 39009085
- [Derived] Allweiss L, Volmari A, Suri V, Wallin JJ, Flaherty JF, Manuilov D, Downie B, Lutgehetmann M, Bockmann JH, Urban S, Wedemeyer H, Dandri M. Blocking viral entry with bulevirtide reduces the number of HDV-infected hepatocytes in human liver biopsies. J Hepatol. 2024 Jun;80(6):882-891. doi: 10.1016/j.jhep.2024.01.035. Epub 2024 Feb 8. PMID 38340811
- [Derived] Hollnberger J, Liu Y, Xu S, Chang S, Martin R, Manhas S, Aeschbacher T, Han B, Yazdi T, May L, Han D, Shornikov A, Flaherty J, Manuilov D, Suri V, Asselah T, Lampertico P, Wedemeyer H, Aleman S, Richards C, Mateo R, Maiorova E, Cihlar T, Mo H, Urban S. No virologic resistance to bulevirtide monotherapy detected in patients through 24 weeks treatment in phase II and III clinical trials for chronic hepatitis delta. J Hepatol. 2023 Sep;79(3):657-665. doi: 10.1016/j.jhep.2023.04.027. Epub 2023 Apr 27. PMID 37120031
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT03852719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany, Italy, Russia, and Sweden.
Pre-assignment Details: 183 participants were screened.
Groups:
- Delayed Treatment/Bulevirtide 10 mg/Day: After an observational period of 48 weeks, participants received bulevirtide 10 mg/day subcutaneous (SC) injection for 96 weeks and were followed for up to 96 weeks (Up to Week 240).
- Bulevirtide 2 mg/Day: Participants received bulevirtide 2 mg/day SC injection for 144 weeks and were followed for up to 96 weeks (Up to Week 240).
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg/day SC injection for 144 weeks and were followed for up to 96 weeks (Up to Week 240).
Period: Overall Study
Arm/Group | Delayed Treatment/Bulevirtide 10 mg/Day | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day
Started | 51 | 49 | 50
Did Not Receive Bulevirtide | 1 | 0 | 0
Completed | 28 | 28 | 30
Not Completed | 23 | 21 | 20
Not completed — Withdrawal of consent | 8 | 8 | 9
Not completed — Physician Decision | 5 | 4 | 1
Not completed — Pregnancy | 2 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Reason not Specified | 3 | 3 | 5
Not completed — Adverse Event | 2 | 1 | 4
Not completed — Progressive disease | 1 | 4 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) included all participants who were randomized to bulevirtide and took at least 1 dose of bulevirtide and those who were randomized to delayed treatment group.
Groups:
- Delayed Treatment/Bulevirtide 10 mg/Day: After an observational period of 48 weeks, participants received bulevirtide 10 mg/day SC injection for 96 weeks and were followed for up to 96 weeks (Up to Week 240).
- Total: Total of all reporting groups
Arm/Group | Delayed Treatment/Bulevirtide 10 mg/Day | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Total
Number analyzed (Participants) | 51 | 49 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 51 | 49 | 50 | 150
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (7.5) | 44 (9.0) | 41 (8.5) | 42 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 19 | 20 | 64
  Male | 26 | 30 | 30 | 86
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 8 | 6 | 25
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1
  White | 40 | 41 | 43 | 124
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 7 | 6 | 14 | 27
  Italy | 7 | 11 | 6 | 24
  Russia | 29 | 28 | 28 | 85
  Sweden | 8 | 4 | 2 | 14
Hepatitis Delta Virus (HDV) Ribonucleic Acid (RNA) [Mean (Standard Deviation); unit: log10 IU/mL] | 5.08 (1.358) | 5.10 (1.194) | 4.96 (1.461) | 5.04 (1.336)
Liver stiffness [Mean (Standard Deviation); unit: kPa] | 15.3 (8.95) | 14.0 (8.19) | 14.8 (9.26) | 14.7 (8.77)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Combined Response at Week 48
Description: Combined response was defined as fulfilment of two conditions simultaneously: Undetectable (< lower limit of quantification (LLOQ, target not detected)) HDV RNA or decrease by ≥ 2 log10 IU/mL from baseline; and ALT normalization.
Time Frame: Week 48
Population: The Full Analysis Set included participants randomized to delayed treatment arm or randomized to bulevirtide and received bulevirtide at least once after randomization. Participants were grouped according to randomized treatment. The arm titles and descriptions in this outcome measure are entered accordingly.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Delayed Treatment: Observation period of 48 weeks.
- Bulevirtide 2 mg/Day: Participants received bulevirtide 2 mg/day SC injection for 48 weeks.
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg/day SC injection for 48 weeks.
Arm/Group | Delayed Treatment | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 51 | 49 | 50
percentage of participants | 2.0 [0.0 to 10.4] | 44.9 [30.7 to 59.8] | 48.0 [33.7 to 62.6]
Statistical Analysis 1: Comparison: Delayed Treatment vs Bulevirtide 10 mg/Day; Test type: Other; p < 0.0001, Fisher Exact — Fisher's exact test was used for comparison of bulevirtide 10 mg versus Delayed Treatment using a significance level of 0.04 at Week 48; Difference in percentages = 46.0, 96% CI 2-sided [30.5 to 61.4]
Statistical Analysis 2: Comparison: Delayed Treatment vs Bulevirtide 2 mg/Day; Test type: Other; p < 0.0001, Fisher Exact — Fisher's exact test was used for comparison of bulevirtide 2 mg versus Delayed Treatment using a significance level of 0.04 at Week 48; Difference in percentages = 42.9, 96% CI 2-sided [27.0 to 58.5]

2. Secondary Outcome: Percentage of Participants With Undetectable HDV RNA at Week 48
Description: Undetectable HDV RNA at Week 48 means undetectable (< LLOQ, target not detected) HDV RNA at Week 48.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed. Participants were grouped according to randomized treatment. The arm titles and descriptions in this outcome measure are entered accordingly.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delayed Treatment | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 51 | 49 | 50
percentage of participants | 0 [0.0 to 7.0] | 12.2 [4.6 to 24.8] | 20.0 [10.0 to 33.7]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.4139, Fisher Exact — Fisher's exact test was used for the comparison of bulevirtide 10 mg versus bulevirtide 2 mg using a significance level of 0.04 at Week 48; Difference in percentages = 7.8, 96% CI 2-sided [-8.5 to 24.3]

3. Secondary Outcome: Percentage of Participants With Alanine Aminotransferase (ALT) Normalization at Week 48
Description: ALT normalization was defined as an ALT value within the normal range, based on the central laboratories [Russian sites: ≤ 31 U/L for females and ≤ 41 U/L for males; all other sites: ≤ 34 U/L for females and ≤ 49 U/L for males])
Time Frame: Week 48
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Delayed Treatment | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 51 | 49 | 50
percentage of participants | 11.8 [4.4 to 23.9] | 51.0 [36.3 to 65.6] | 56.0 [41.3 to 70.0]
Statistical Analysis 1: Comparison: Delayed Treatment vs Bulevirtide 2 mg/Day; Test type: Other; p < 0.0001, Fisher Exact — Fisher's exact test was used for comparison of bulevirtide 2 mg versus Delayed treatment using a significance level of 0.05; Difference in percentages = 39.3, 95% CI 2-sided [20.0 to 55.8]
Statistical Analysis 2: Comparison: Delayed Treatment vs Bulevirtide 10 mg/Day; Test type: Other; p < 0.0001, Fisher Exact — Fisher's exact test was used for comparison of bulevirtide 10 mg versus Delayed treatment using a significance level of 0.05; Difference in percentage = 44.2, 95% CI 2-sided [25.8 to 59.9]

4. Secondary Outcome: Change From Baseline in Liver Stiffness, as Measured by Elastography at Week 48
Description: ANCOVA was used for analysis.
Time Frame: Baseline (Baseline for Delayed Treatment/Bulevirtide 10 mg/day is reset at Week 48), Week 48
Population: Participants in the Full Analysis Set with available data were analyzed. Data is reported separately for changes from Baseline at Week 48 for the Delayed Treatment arm and for Delayed Treatment/Bulevirtide 10 mg/day arm after 48 weeks of bulevirtide 10 mg treatment. Participants were grouped according to randomized treatment and study design. The arm titles and descriptions in the outcome measure are entered accordingly.
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Groups:
- Delayed Treatment / /Bulevirtide 10 mg/Day: Participants received Bulevirtide 10 mg/Day SC for 48 weeks after an observation period of 48 weeks.
Arm/Group | Delayed Treatment | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment / /Bulevirtide 10 mg/Day
Number analyzed (Participants) | 46 | 48 | 42 | 48
kPa | 0.87 [-0.79 to 2.53] | -3.06 [-4.67 to -1.45] | -3.16 [-4.88 to -1.43] | -3.36 [-4.60 to -2.12]
Statistical Analysis 1: Comparison: Delayed Treatment vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.0010, ANCOVA; Difference in LS Mean = -4.02, 95% CI 2-sided [-6.39 to -1.65]
Statistical Analysis 2: Comparison: Delayed Treatment vs Bulevirtide 2 mg/Day; Test type: Other; p = 0.0009, ANCOVA; Difference in LS Mean = -3.93, 95% CI 2-sided [-6.23 to -1.63]

5. Secondary Outcome: Change From Baseline in Liver Stiffness, as Measured by Elastography at Week 96
Description: Mixed model for repeated measurements (MMRM) was used for analysis.
Time Frame: Baseline (Baseline for Delayed Treatment/Bulevirtide 10 mg/day is reset at Week 48), Week 96
Population: Participants from Full Analysis Set with available data were analyzed. Participants were grouped according to randomized treatment and study design. The arm titles and descriptions in the outcome measure are entered accordingly.
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Groups:
- Bulevirtide 2 mg/Day: Participants received bulevirtide 2 mg/day SC injection for 96 weeks which continued up to 144 weeks and were followed for 96 weeks (Up to Week 240).
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg/day SC injection for 96 weeks which continued up to 144 weeks and were followed for 96 weeks (Up to Week 240).
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment/Bulevirtide 10 mg/Day
Number analyzed (Participants) | 47 | 47 | 48
kPa | -4.31 [-5.54 to -3.08] | -4.88 [-6.11 to -3.65] | -4.20 [-5.41 to -2.98]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.5156, MMRM; Difference in Least Square (LS) Mean = 0.57, 95% CI 2-sided [-1.16 to 2.30]

6. Secondary Outcome: Change From Baseline in Liver Stiffness, as Measured by Elastography at Week 144
Description: MMRM was used for analysis.
Time Frame: Baseline, Week 144
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Groups:
- Bulevirtide 2 mg/Day: Participants received bulevirtide 2 mg/day SC for 144 weeks and were followed for up to 96 weeks (Up to Week 240).
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day
Number analyzed (Participants) | 45 | 43
kPa | -5.24 [-6.85 to -3.63] | -4.03 [-5.67 to -2.40]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Other; p = 0.2977, MMRM; Difference in Least Square (LS) Mean = -1.21, 95% CI 2-sided [-3.50 to 1.08]

7. Secondary Outcome: Change From Baseline in Liver Stiffness, as Measured by Elastography at Week 192
Description: MMRM was used for analysis.
Time Frame: Baseline (Baseline for Delayed Treatment/Bulevirtide 10 mg/day is reset at Week 48), Week 192
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment/Bulevirtide 10 mg/Day
Number analyzed (Participants) | 35 | 34 | 35
kPa | -3.74 [-5.28 to -2.20] | -3.70 [-5.27 to -2.14] | -1.91 [-3.49 to -0.34]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Superiority; p = 0.9719, MMRM — P-value was based on the mixed-effects model for repeated measurements (MMRM) model; LS-Mean of Diffrence = -0.04, 95% CI 2-sided [-2.23 to 2.15] — Least squares (LS) means, standard errors (SE), 95% CIs and p-values were based on the mixed-effects model for repeated measurements (MMRM) model for change from baseline

8. Secondary Outcome: Change From Baseline in Liver Stiffness, as Measured by Elastography at Week 240
Description: MMRM was used for analysis.
Time Frame: Baseline (Baseline for Delayed Treatment/Bulevirtide 10 mg/day is reset at Week 48), Week 240
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: kPa
Groups:
- Delayed Treatment/ Bulevirtide 10 mg/Day: After an observational period of 48 weeks, participants received bulevirtide 10 mg/day SC injection for 96 weeks and were followed for up to 96 weeks (Up to Week 240).
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment/ Bulevirtide 10 mg/Day
Number analyzed (Participants) | 28 | 29 | 28
kPa | -1.20 [-3.71 to 1.31] | -3.31 [-5.78 to -0.84] | -3.59 [-6.14 to -1.04]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Superiority — P-value was based on the mixed-effects model for repeated measurements (MMRM) model; p = 0.2369, MMRM; LS-Mean of Difference = 2.11, 95% CI 2-sided [-1.41 to 5.63] — [estimate comment as in outcome 7, analysis 1]

9. Secondary Outcome: Percentage of Participants With Undetectable HDV RNA 24 Weeks After Scheduled End of Treatment (Sustained Virological Response)
Description: Undetectable HDV RNA 24 Weeks after Scheduled End of Treatment means undetectable (< LLOQ, target not detected) HDV RNA at Week 168
Time Frame: Week 168
Population: Participants in the Full Analysis Set were analyzed. Participants were grouped according to randomized treatment and study design. The arm titles and descriptions in the outcome measure are entered accordingly.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment/Bulevirtide 10 mg/Day
Number analyzed (Participants) | 49 | 50 | 50
percentage of participants | 18.4 [8.8 to 32.0] | 26.0 [14.6 to 40.3] | 18.0 [8.6 to 31.4]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Superiority; p = 0.4695, Fisher Exact — P-value was based on Fisher's Exact Test; Response Rate Difference = 7.6, 95% CI 2-sided [-9.6 to 24.4] — For response rate difference, the 95% exact unconditional confidence interval (CI) based on the score statistic was presented
Statistical Analysis 2: Comparison: Bulevirtide 2 mg/Day vs Delayed Treatment/Bulevirtide 10 mg/Day; Test type: Superiority; p = 1.0000, Fisher Exact — P-value was based on Fisher's Exact Test; Response Rate Difference = -0.4, 95% CI 2-sided [-16.3 to 15.5] — [estimate comment as in outcome 9, analysis 1]

10. Secondary Outcome: Percentage of Participants With Undetectable HDV RNA 48 Weeks After Scheduled End of Treatment (Sustained Virological Response)
Description: Undetectable HDV RNA 48 Weeks after Scheduled End of Treatment means undetectable (< LLOQ, target not detected) HDV RNA at Week 192
Time Frame: Week 192
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment/Bulevirtide 10 mg/Day
Number analyzed (Participants) | 49 | 50 | 50
percentage of participants | 16.3 [7.3 to 29.7] | 24.0 [13.1 to 38.2] | 16.0 [7.2 to 29.1]
Statistical Analysis 1: Comparison: Bulevirtide 2 mg/Day vs Bulevirtide 10 mg/Day; Test type: Superiority; p = 0.4539, Fisher Exact — P-value was based on Fisher's Exact Test; Response Rate Difference = 7.7, 95% CI 2-sided [-8.8 to 24.0] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Bulevirtide 2 mg/Day vs Delayed Treatment/Bulevirtide 10 mg/Day; Test type: Superiority; p = 1.0000, Fisher Exact — P-value was based on Fisher's Exact Test; Response Rate Difference = -0.3, 95% CI 2-sided [-15.6 to 15.5] — [estimate comment as in outcome 9, analysis 1]

11. Secondary Outcome: Percentage of Participants Who Prematurely Discontinued Study Drug Due to an Adverse Event (AE) by Week 144
Description: An AE was defined as any untoward medical occurrence in a participant administered study drug and which did not necessarily have a causal relationship with the study drug. An AE could therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study drug, whether or not related to the study drug.
Time Frame: Delayed Treatment/Bulevirtide 10 mg/day arm: Week 48 up to Week 144; Bulevirtide 2mg/day and 10 mg/day arms: First dose date up to Week 144
Population: Participants in the SAS were analyzed. The SAS included all participants who were randomized into the study and took at least 1 dose of bulevirtide study drug, or who were randomized to the delayed treatment group. Participants were grouped according to actual treatment received for time points Week 0 to 144. The arm titles and descriptions in this outcome measure are entered accordingly.
Measure: Number; unit: percentage of participants
Groups:
- Bulevirtide 2 mg/Day: Participants received bulevirtide 2 mg/day SC injection for 144 weeks.
- Bulevirtide 10 mg/Day: Participants received bulevirtide 10 mg/day SC injection for 144 weeks.
- Delayed Treatment/Bulevirtide 10 mg/Day: After an observational period of 48 weeks, participants received bulevirtide 10 mg/day SC injection for 96 weeks.
Arm/Group | Bulevirtide 2 mg/Day | Bulevirtide 10 mg/Day | Delayed Treatment/Bulevirtide 10 mg/Day
Number analyzed (Participants) | 49 | 50 | 50
percentage of participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Up to Week 240; Adverse Events: Up to Week 48 (first 3 arms); Up to Week 144 (arms 4 and 5); Up to Weeks 48-144 (arm 6); >Week 144 up to Week 240 (arms 7-9). Adverse Event: SAS included all participants randomized (posttreatment SAS required >=1 measurement after EOT) delayed treatment arm or randomized to bulevirtide and received bulevirtide at least once after randomization. All-cause mortality: Randomized Set included all enrolled and randomized participants.
Description: Participants were grouped according to actual treatment received for time points Week (Wk) 0 to 48, 0 to 144, Wk 48 to 144 and by last treatment received after Wk 144, up to Wk 240. The arm titles and descriptions in this section are entered accordingly. Actual treatment received is defined as randomized treatment except for participants who received treatment that differs from randomized treatment for the entire treatment duration.
Groups:
- Delayed Treatment (Baseline to Week 48): Observation for 48 weeks.
- Bulevirtide 2 mg/Day (Baseline to Week 48): Bulevirtide 2 mg/day SC for 48 weeks.
- Bulevirtide 10 mg/Day (Baseline to Week 48): Bulevirtide 10 mg/day SC for 48 weeks.
- Bulevirtide 2 mg/Day (Baseline to Week 144): Participants received bulevirtide 2 mg/day SC for 144 weeks.
- Bulevirtide 10 mg/Day (Baseline to Week 144): Participants received bulevirtide 10 mg/day SC for 144 weeks.
- Delayed Treatment/Bulevirtide 10 mg/Day (Week 48 to Week 144): After an observational period of 48 weeks, participants received bulevirtide 10 mg/day SC for 96 weeks (Up to Week 144).
- Bulevirtide 2 mg/Day (After EOT (>Week 144 up to Week 240)): After 144 weeks of treatment with bulevirtide 2 mg/day SC, participants were followed for up to 96 weeks (Up to Week 240).
- Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240): After 144 weeks of treatment with bulevirtide 10 mg/day SC, participants were followed for up to 96 weeks (Up to Week 240).
- Delayed Treatment/Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240): After 96 weeks of treatment (Up to Week 144) with bulevirtide 10 mg/day SC, participants were followed for up to 96 weeks (Up to Week 240).
Arm/Group | Delayed Treatment (Baseline to Week 48) | Bulevirtide 2 mg/Day (Baseline to Week 48) | Bulevirtide 10 mg/Day (Baseline to Week 48) | Bulevirtide 2 mg/Day (Baseline to Week 144) | Bulevirtide 10 mg/Day (Baseline to Week 144) | Delayed Treatment/Bulevirtide 10 mg/Day (Week 48 to Week 144) | Bulevirtide 2 mg/Day (After EOT (>Week 144 up to Week 240)) | Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240) | Delayed Treatment/Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240)
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49 | 0/50 | 0/49 | 0/50 | 1/50 | 0/46 | 0/47 | 0/49
Serious Adverse Events (participants affected / at risk) | 1/51 | 2/49 | 1/50 | 3/49 | 6/50 | 3/50 | 7/46 | 7/47 | 8/49
Other Adverse Events (participants affected / at risk) | 30/51 | 35/49 | 41/50 | 44/49 | 46/50 | 41/50 | 31/46 | 33/47 | 34/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Delayed Treatment (Baseline to Week 48) (N=51) | Bulevirtide 2 mg/Day (Baseline to Week 48) (N=49) | Bulevirtide 10 mg/Day (Baseline to Week 48) (N=50) | Bulevirtide 2 mg/Day (Baseline to Week 144) (N=49) | Bulevirtide 10 mg/Day (Baseline to Week 144) (N=50) | Delayed Treatment/Bulevirtide 10 mg/Day (Week 48 to Week 144) (N=50) | Bulevirtide 2 mg/Day (After EOT (>Week 144 up to Week 240)) (N=46) | Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240) (N=47) | Delayed Treatment/Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240) (N=49)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Varices oesophageal (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic hepatitis B (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coronavirus pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Covid-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hepatitis D (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 2
Hepatitis E (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Yersinia infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Delayed Treatment (Baseline to Week 48) (N=51) | Bulevirtide 2 mg/Day (Baseline to Week 48) (N=49) | Bulevirtide 10 mg/Day (Baseline to Week 48) (N=50) | Bulevirtide 2 mg/Day (Baseline to Week 144) (N=49) | Bulevirtide 10 mg/Day (Baseline to Week 144) (N=50) | Delayed Treatment/Bulevirtide 10 mg/Day (Week 48 to Week 144) (N=50) | Bulevirtide 2 mg/Day (After EOT (>Week 144 up to Week 240)) (N=46) | Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240) (N=47) | Delayed Treatment/Bulevirtide 10 mg/Day (After EOT (>Week 144 up to Week 240) (N=49)
Anaemia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 5 | 3 | 3 | 1 | 1 | 5
Eosinophilia (Blood and lymphatic system disorders) | 0 | 5 | 5 | 5 | 5 | 1 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 10 | 7 | 5 | 10 | 9 | 7 | 2 | 4 | 5
Lymphopenia (Blood and lymphatic system disorders) | 4 | 4 | 4 | 8 | 6 | 5 | 3 | 4 | 7
Neutropenia (Blood and lymphatic system disorders) | 3 | 2 | 5 | 8 | 10 | 3 | 3 | 4 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 5 | 5 | 10 | 8 | 7 | 6 | 5 | 7
Bradycardia (Cardiac disorders) | 0 | 0 | 3 | 1 | 3 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 2 | 3 | 4 | 1 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 4 | 2 | 4 | 2 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 5 | 2 | 5 | 2 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 3 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 4 | 3 | 6 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 2 | 2 | 2 | 1 | 3 | 4 | 4
Fatigue (General disorders) | 1 | 5 | 7 | 7 | 9 | 3 | 0 | 5 | 4
Injection site erythema (General disorders) | 0 | 2 | 5 | 3 | 5 | 2 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 2 | 3 | 2 | 3 | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 0 | 3 | 5 | 3 | 6 | 3 | 0 | 0 | 0
Injection site swelling (General disorders) | 0 | 1 | 3 | 1 | 3 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 2 | 0 | 3 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 3 | 4 | 1 | 1 | 2 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 5 | 4 | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2 | 2 | 4 | 2 | 3 | 1 | 0 | 1
Covid-19 (Infections and infestations) | 1 | 1 | 0 | 5 | 8 | 5 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 4 | 0 | 5 | 2 | 3 | 2 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 2 | 2 | 6 | 2 | 1 | 2 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 0 | 1 | 0 | 1 | 2 | 2 | 3 | 1
Alanine aminotransferase increased (Investigations) | 4 | 2 | 3 | 5 | 4 | 0 | 19 | 11 | 18
Alpha-2 macroglobulin increased (Investigations) | 1 | 0 | 0 | 4 | 3 | 2 | 2 | 3 | 6
Amylase increased (Investigations) | 1 | 1 | 0 | 3 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 1 | 2 | 1 | 1 | 17 | 11 | 15
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 2 | 1 | 3 | 1 | 0 | 2 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 2 | 1 | 3 | 2 | 8 | 4 | 3
Hepatitis D RNA positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0
Lipase increased (Investigations) | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 2 | 0
Transaminases increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 7 | 2
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 13 | 7 | 7 | 22 | 19 | 14 | 6 | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4 | 6 | 8 | 1 | 2 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 1 | 3 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 2 | 3 | 2 | 4 | 1 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 9 | 10 | 10 | 12 | 7 | 0 | 1 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 3 | 0 | 3 | 0 | 0 | 2 | 0
Proteinuria (Renal and urinary disorders) | 2 | 3 | 1 | 4 | 3 | 2 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 2 | 3 | 3 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 6 | 7 | 6 | 8 | 0 | 1 | 3 | 1
Hypertension (Vascular disorders) | 0 | 1 | 3 | 3 | 4 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (7):
  • Study Protocol: Amendment 4 (2022-04-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/Prot_000.pdf
  • Study Protocol: Amendment 6 (2023-01-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/Prot_002.pdf
  • Statistical Analysis Plan: Week 48 Analysis (2021-08-20): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/SAP_001.pdf
  • Statistical Analysis Plan: Week 96 Analysis (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/SAP_003.pdf
  • Statistical Analysis Plan: Week 144 Analysis (2023-06-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/SAP_004.pdf
  • Statistical Analysis Plan: Week 192 Analysis (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/SAP_005.pdf
  • Statistical Analysis Plan: Statistical Analysis Plan: Week 240 Analysis (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03852719/SAP_006.pdf